CLINICAL TRIAL: NCT05209282
Title: The Effect Of Video Based Action Observation Training And Live Action Observation Training On Motor Function, Activity Participation And Secondary Outcome Measures İn Children With Spastic Diplegic Cerebral Palsy
Brief Title: Diplegic Cerebral Palsy and Action Observation Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Inonu University (Other)
Responsible Party: Principal Investigator, Burcu Talu, Assoc., Inonu University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2021/2663
Record Dates: First submitted 2022-01-13; First posted 2022-01-26 (Actual); Last update posted 2024-02-09 (Actual); Status verified 2023-04

CONDITIONS: Diplegic Cerebral Palsy
Keywords: Action Observation Therapy; Diplegic Cerebral Palsy; Mirror Neuron System; Motor Function; Activity Participation; Secondary Outcome Measures
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Intervention Model Description: Experimental, Randomized Controlled Study
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Grup I (Experimental): Conventional physiotherapy program, Video-based action observation training
  Interventions: Other: Video Based Action Observation; Other: Conventional physiotherapy program
- Grup II (Experimental): Conventional physiotherapy program, Live Action Observation Training
  Interventions: Other: Live Action Observation; Other: Conventional physiotherapy program
- Grup III (Other): Conventional physiotherapy program
  Interventions: Other: Conventional physiotherapy program

INTERVENTIONS:
Other: Video Based Action Observation — Individuals in this group will receive video-based action observation training in addition to the conventional physiotherapy program.
  Other Names: Conventional physiotherapy program
  Arms: Grup I
Other: Live Action Observation — Individuals in this group will receive live action observation training in addition to the conventional physiotherapy program.
  Other Names: Conventional physiotherapy program
  Arms: Grup II
Other: Conventional physiotherapy program — Individuals in this group will only receive a conventional physiotherapy program.

SUMMARY:
In this study, video-based action observation training and live action observation training in children with spastic diplegic cerebral palsy; It was aimed to examine the effect on motor function, activity participation and secondary outcome measures.

DETAILED DESCRIPTION:
The study was designed as a single-blind randomized controlled trial. Patients aged 5-14 years with spastic diplegic cerebral palsy will be included. Children will be assigned to groups through stratified randomisation; The patients will be divided into 3 groups as experimental and control groups. Group 1 (experiment): video-based action observation training in addition to the conventional rehabilitation program, Group 2 (experiment): live action observation training in addition to the conventional rehabilitation program, Group 3 (control) will receive only the conventional rehabilitation program. The experimental group will receive 20 minutes of action observation training after a conventional physiotherapy program for 20 minutes for 8 weeks, 40 minutes 2 days a week. The control group will receive 40 minutes of conventional treatment. Evaluations will be made for each group, before and 8 weeks after the start of the study. GMFM for gross motor function; Pediatric berg balance scale for balance function; Timed Up and Go Test for functional mobility assessment; Gillette Functional Assessment Questionnaire and 1-min walk test to assess functional walking; sit and stand test for functional muscle strength and to evaluate activity participation; The Child and Adolescent Participation Questionnaire (CASP) will be used.

ELIGIBILITY:
Inclusion Criteria:

* Being diagnosed with spastic diplegic cerebral palsy,
* To be between the ages of 5-14,
* To be at GMFCS I, II and III levels,
* To have the cognitive level to follow the instructions given by the researchers,
* IQ> 70 (to be accessed from patient files),
* Those who do not have serious restrictions in joint movement,

Exclusion Criteria:

* Children with joint contractures,
* Not having visual impairment and visual field defect,
* Children who have had a seizure in the last 6 months or children who cannot be controlled despite seizure medication
* Those who received botulinum injections 6 months before the study.

Ages: 5 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 39 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-02-24 (Actual); Study Completion 2022-10-31 (Actual)

PRIMARY OUTCOMES:
Gross Motor Function Measure | 8weeks
  Gross Motor Function measure is used to evaluate Motor Functions
The Child and Adolescent Scale of Participation (CASP) | 8weeks
  The CASP questionnaire is a questionnaire that evaluates the individual's community participation in the home, school, neighborhood settings.

SECONDARY OUTCOMES:
Pediatric berg balance scale | 8weeks
  The test is performed progressively from timed sitting balance to standing on one leg.
Timed Up and Go Test (TUG) | 8weeks
  It is a test that measures the mobility of the child and evaluates both dynamic and static balance.
Gillette Functional Assessment Questionnaire | 8weeks
  Gillette FDA is a self-reported or self-reported assessment. Gillette FDA; It includes the FDA Gait Scale, which classifies ambulation function at 10 levels, and the 22-item Skills Test assessing functional locomotor activity.
One-Minute Walk Test | 8weeks
  It is an inexpensive and user-friendly test that can be used to assess functional ability with the 1-minute fast walking test. During the test, children wear their comfortable clothes and shoes. Children who wear orthoses are evaluated with orthoses, and children who walk with a mobility aid are evaluated with mobility aids.
Sit to Stand Test | 8weeks
  The child is asked to get up from a chair without armrests and sit back down again, with his hips and knees flexed to 90 degrees and his feet in full contact with the ground. The time to sit and stand up to 5 times is determined by the stopwatch.

CONTACTS AND LOCATIONS:
Overall Officials: Burcu TALU, Assoc. Prof., Principal Investigator — Inonu University
Locations (1):
- Inonu University, Malatya, Battalgazi/MALATYA, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No